CLINICAL TRIAL: NCT07365527
Title: Tumor Response to Sonoporation: A Clinical Translational RCT of Contrast-enhanced Ultrasound Induced Changes in Tumor Microenvironment of Colorectal Liver Metastases
Brief Title: Sonoporation and Tumor Microenvironment Response in Colorectal Liver Metastases
Acronym: CEUSON
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ismail Gögenur, Professor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-2025-19453
Record Dates: First submitted 2025-12-19; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Liver Metastases From Colorectal Cancer
Keywords: liver metastasis; CEUS; Sonoporation; Contrast enhanced ultrasound; colorectal cancer; liver metastases; tumor microenvironment
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients in the intervention group will be randomized to receive either high-intensity CEUS or low-intensity CEUS. Patients in the intervention group will be compared to a historical control group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Historical control group (No Intervention): The historical control group consists of 24 matched patients who underwent liver resection for one or more colorectal liver metastases at Rigshospitalet between 2022 and the end of 2024. These patients serve as a non-intervention comparison cohort.
- Low-intensity CEUS intervention group (Experimental): 12 eligible patients will be randomized to receive LI-CEUS intervention
  Interventions: Other: Low-intensity contrast enhanced ultrasound
- High-intensity CEUS intervention group (Experimental): 12 eligible patients will be randomized to receive HI-CEUS intervention
  Interventions: Other: High-intensity contrast enhanced ultrasound

INTERVENTIONS:
Other: Low-intensity contrast enhanced ultrasound — The LI-CEUS arm will receive a 30-minute contrast-enhanced ultrasound session targeting a designated study metastasis. During the procedure, 1 mL of the ultrasound contrast agent SonoVue will be administered every 3 minutes throughout the entire session. Minimum 7 days after the intervention a biopsy of the study metastasis will be conducted.
  Arms: Low-intensity CEUS intervention group
Other: High-intensity contrast enhanced ultrasound — The HI-CEUS intervention group will recieve a 30-minute CEUS procedure targeting a designated study metastasis. During the procedure, 1 mL of the ultrasound contrast agent SonoVue will be administered every 3 minutes throughout the entire session. A high-intensity ultrasound "flash" will be applied every 30 seconds. This "flash" consists of a brief sequence of ultrasound waves with a high mechanical index that causes complete destruction of microbubbles within the imaging field. Minimum 7 days after the intervention a biopsy of the study metastasis will be conducted.
  Arms: High-intensity CEUS intervention group

SUMMARY:
This study is an investigator-initiated, randomized controlled trial enrolling patients with colorectal liver metastases. The objectives are to evaluate the safety and efficacy of contrast-enhanced ultrasound (CEUS)-mediated sonoporation as a potential therapeutic intervention and to investigate whether sonoporation can modulate the tumor microenvironment toward a more immune-active state

DETAILED DESCRIPTION:
The trial is designed as an investigator-initiated, multicenter, prospective, randomized, controlled, two-arm, intervention trial with a matched historical control group aims to evaluate the therapeutic potential of contrast-enhanced ultrasound (CEUS) in patients with colorectal liver metastases (CLM). The primary objectives are to assess whether CEUS can modulate the tumor microenvironment and to determine the safety, tolerability, and feasibility of CEUS as a therapeutic modality. Eligible patients will be randomized to receive either low-intensity CEUS (LI-CEUS) or high-intensity CEUS (HI-CEUS) focused on a designated study metastasis. Safety, feasibility, and success-rate of the intervention will be registered. Minimum seven days post-intervention a biopsy of the study metastasis will be conducted. Subsequent analyses will compare immune cell infiltration, immune-related gene expression, and stromal and vascular remodeling in LI-CEUS- and HI-CEUS-exposed metastases versus historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Ability to provide written informed consent
* Histopathological confirmed colorectal adenocarcinoma
* Scheduled for liver resection or ablation at the Rigshospital, or admitted to oncologic treatment due to colorectal liver metastases (CLM) at Zealand University Hospital
* Presence of at least one CLM evaluable and accessible by CEUS
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Follow the conditions regarding fertility, pregnancy, or lactation:

  * Women of childbearing potential (WOCBP) are defined as women ranging from the period of menarche till the post-menopausal period, unless permanently sterile (e.g. hysterectomy, bilateral salpingectomy and bilateral oophorectomy), Post-menopause is defined as no menses for 12 months without an alternative medical cause.
  * WOCBP should use a secure and highly effective birth control (as stated in the "Recommendations related to contraception and pregnancy testing in clinical trials", version 1.1, section 4.1, from the Clinical Trials Facilitation and Coordination Group) during the entire period of the trial. In cases of uncertainty regarding pregnancy, pregnancy testing either as highly sensitive serum or urine pregnancy test will be used.

Exclusion Criteria:

* Oncologic systemic treatment 2 weeks prior to inclusion
* Prior treatment with an immune checkpoint inhibitor (e.g. anti-PD-L1, anti PD-1, or anti-PD-L2)
* Inability to reliably distinguish the study metastasis from other hepatic metastases using CEUS
* Systemic treatment with either corticosteroids (>10 mg daily prednisolone equivalents) or other immunosuppressive medications within 2 weeks prior inclusion. Inhaled or topical steroids and adrenal replacements doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Known history of human immunodeficiency virus (HIV), active or chronic hepatitis B, or C.
* Pregnancy or lactation.
* Confirmed dMMR positive primary tumors
* Inability to comply with study protocol due to psychological, social, or logistical reasons.
* Contraindications for CEUS:

  * Known hypersensitivity to SonoVue® or any other ultrasound contrast agent
  * Uncontrolled atrial hypertension
  * Known right-to-left intracardiac shunt
  * Severe pulmonary hypertension (SAP >90 mmHg)
  * Adult respiratory distress syndrome.
  * Known hypersensitivity to macrogols
  * Unstable ischemic heart disease or acute coronary syndrome
  * Severe lung disease, e.g. severe chronic obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Immune cell density (CD8+, CD3+) in colorectal liver metastases exposed to LI-CEUS or HI-CEUS, compared to controls. | ≥7 days after postinterventional

SECONDARY OUTCOMES:
Number of participants in the intervention group with treatment-related adverse events assessed by CTCAE v5.0 | Daily, until 7 days post-interventional
Procedure success of LI-CEUS and HI-CEUS procedures as assessed by operator-defined completion of the planned intervention | Periinterventional
Differential expression of immune-related genes between CEUS-exposed and control liver metastases | ≥7 days postinterventional
  Tissue bulk transcriptional analyses will be evaluated by the Nanostring nCounter platform. Immune-related spatial protein profiling of tumor regions will be evaluated by the GeoMx digital spatial profiler
Systemic immune response assessed by changes in the circulating cytokine profiles following LI-CEUS and HI-CEUS | Pre- and ≥7 days postinterventional
Frequency and type of technical issues encountered during LI-CEUS and HI-CEUS procedures assessed by the operator | Periinterventional

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Nolsøe, Professor, Principal Investigator — Center of Surgical Ultrasound, Surgical department of Zealand University Hospital; Ismail Gögenur, Professor, Study Director — Center of Surgical Science, Surgical department of Zealand University Hospital
Locations (1):
- Surgical Department, Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No
It is not yet decided.